CLINICAL TRIAL: NCT01636557
Title: A Phase I, Open-label, Drug Interaction Study to Evaluate the Effect of a Single-dose of CNTO 136 (Sirukumab) on CYP450 Enzyme Activities After Subcutaneous Administration in Subjects With Rheumatoid Arthritis
Brief Title: A Study to Evaluate the Effect of a Single Dose of CNTO 136 (Sirukumab) on CYP450 Enzyme Activities After Subcutaneous Administration in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR100842; CNTO136ARA1001 (Other: Janssen Research & Development, LLC); 2011-001704-35 (EudraCT Number)
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid arthritis; sirukumab; CNTO 136; CYP450 enzyme; anti-interleukin-6 monoclonal antibody
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sirukumab; Midazolam; Warfarin; Vitamin K; Omeprazole; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sirukumab and 5-probe cocktail (Experimental): The 5-probe cocktail will consist of oral doses of midazolam, warfarin/vitamin K, omeprazole, and caffeine.
  Interventions: Drug: Sirukumab; Drug: Midazolam; Drug: Warfarin; Drug: Vitamin K; Drug: Omeprazole; Drug: Caffeine

INTERVENTIONS:
Drug: Sirukumab — Type=exact number, unit=mg, number=300, form=solution for injection, route=subcutaneous use, on Day 8
Drug: Midazolam — Type=exact number, unit=mg/kg, number 0.03, form=commercially available form, route=oral use, on Days 1, 15, 29, and 50
Drug: Warfarin — Type=exact number, unit=mg, number= 10, form=commercially available form, route=oral use, on Days 1, 15, 29, and 50
Drug: Vitamin K — Type=exact number, unit=mg, number =10, form=commercially available form, route=oral use, on Days 1, 15, 29, and 50
Drug: Omeprazole — Type=exact number, unit=mg, number=20, form=commercially available form, route=oral use, on Days 1, 15, 29, and 50
Drug: Caffeine — Type=exact number, unit=mg, number=100, form=commercially available form, route=oral use, on Days 1, 15, 29, and 50

SUMMARY:
The main purpose of this study is to evaluate the potential effects of a single dose of sirukumab on the pharmacokinetics (what the body does to a drug) of study agents that are specific for cytochrome P450 (CYP) enzymes (CYP3A4, CYP2C9, CYP2C19, and CYP1A2) in patients with active rheumatoid arthritis (RA). This study will also assess the safety and tolerability of a single subcutaneous (SC, under the skin) dose of sirukumab in patients with active RA.

DETAILED DESCRIPTION:
This is an open-label (all patients and study personnel will know the identity of the administered study agents), multi-center, drug-drug interaction study. Approximately 18 patients may be enrolled in this study, and there will be one treatment group. All patients will receive a single subcutaneous (SC) dose of sirukumab. Cytochrome P450 (CYP) enzyme-specific study agents (5-probe cocktail) will consist of oral doses of midazolam, warfarin/vitamin K, omeprazole, and caffeine administered on 4 separate occasions throughout the study. A blood sample for CYP genetic analysis (genotyping) will be collected during screening from all prospective patients to determine eligibility for the study. Participation in CYP genotyping prescreening is mandatory for all patients. The CYP genotyping blood sample will not be used for any additional genetic research and will be destroyed after completion of this study. The total duration of study participation will be approximately 12 weeks for all patients included in the study, including a screening visit up to 4 weeks prior to first study agent administration. Patients will have five in-patient periods, four consisting of 3 days and 2 nights each and one consisting of 2 days and 1 night. Patients safety will be monitored throughout the study, and there will be approximately 7 weeks of safety follow-up after sirukumab administration.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index of 18 kg/m2 to 29.9 kg/m2, inclusive, and a body weight of 60 kg to 110 kg, inclusive, if a man, and 50 kg to 100 kg, inclusive, if a woman
* Have a diagnosis of rheumatoid arthritis (RA) for at least 3 months before screening
* If using nonsteroidal anti-inflammatory drugs (NSAIDs) or other analgesics, must be on a stable dose for at least 2 weeks prior to Day 1 (use of indomethacin is excluded)
* If using methotrexate (MTX), sulfasalazine, hydroxychloroquine, chloroquine, or bucillamine, should have started treatment at least 3 months prior to Day 1, have no serious toxic side effects attributable to these agents, and be on a stable dose for at least 4 weeks prior to Day 1 and remain so during the entire duration of the study. If using MTX, the recommended doses are within the range of 7.5 mg to 25 mg oral or subcutaneous weekly. If currently not using MTX, sulfasalazine, hydroxychloroquine, chloroquine, or bucillamine, must have not received these agents for at least 4 weeks prior to Day 1.
* If using oral corticosteroids, must be on a stable dose equivalent to ≤ 10 mg/day of prednisone for at least 2 weeks prior to Day 1. If currently not using oral corticosteroids, the patient must have not received oral corticosteroids for at least 2 weeks prior to screening

Exclusion Criteria:

* Have received anti-tumor necrosis factor (TNF) agents (eg, infliximab, golimumab, adalimumab, etanercept, or certolizumab pegol) within 3 months of Day 1
* Have a history of tocilizumab (anti-IL-6 receptor) or sirukumab use; have used B-cell depleting therapy (eg, rituximab) within 7 months of Day 1; have used anakinra within 4 weeks of Day 1; have used any other biologic therapy for the treatment of RA within 3 months of Day 1
* Have received intra-articular (IA), intramuscular (IM), intravenous (IV), or topical corticosteroids, including adrenocorticotrophic hormone, during the 4 weeks prior to Day 1
* Have received leflunomide within 24 months of Day 1 and have not undergone a drug elimination procedure, unless the M1 metabolite is measured and is undetectable
* Have a history of cyclophosphamide or cytotoxic agent use; have received cyclosporine A, azathioprine, tacrolimus, mycophenolate mofetil, oral or parenteral gold, D-penicillamine, or IL-1ra (anakinra) within 4 weeks of Day 1; have received an investigational drug (including investigational vaccines) or used an investigational medical device within 3 months or 5 half-lives, whichever is longer, before Day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10-11 (Actual); Primary Completion 2013-10-19 (Actual); Study Completion 2013-10-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of midazolam, S-warfarin, omeprazole, and caffeine | Up to 54 days
  Pharmacokinetic parameters will include the maximum observed plasma concentration (Cmax), time to reach the maximum observed plasma concentration (Tmax), area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration (AUClast), area under the plasma concentration-time curve from time 0 to 96 hours (AUC0-96h) (S-warfarin only), area under the plasma concentration versus time curve from time 0 to infinity with extrapolation of the terminal phase (AUCinf).

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 12 weeks
Clinical laboratory assessments | Up to 12 weeks
  Blood and urine tests
Electrocardiograms (ECGs) | Up to 12 weeks
Vital signs evaluations | Up to 12 weeks
Physical examination | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- Germany (2):
  - Berlin
  - Munich
- Chisinau, Moldova
- Bloemfontein, South Africa
- Seoul, South Korea